CLINICAL TRIAL: NCT00125814
Title: Multi-Center Trial to Evaluate the Efficacy and Safety of Structured Treatment Interruptions With or Without Pegylated Interferon Alpha for HIV-Infected Patients After Prolonged Viral Suppression (ANRS 105 INTERVAC)
Brief Title: Structured Treatment Interruptions With or Without Pegylated Interferon Alpha for HIV-Infected Patients After Prolonged Viral Suppression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 105 INTERVAC
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2005-08-16 (Estimated); Status verified 2005-08

CONDITIONS: HIV Infections
Keywords: Interferon Alfa-2b; HIV infections
MeSH Terms: conditions — HIV Infections | interventions — Interferon alpha-2

INTERVENTIONS:
Drug: Interferon alfa-2b
Procedure: Structured treatment interruptions

SUMMARY:
The purpose of this study is to determine whether the adjunctional of interferon alfa to structured treatment interruptions correlated with a long time off treatment in HIV-1 infection.

DETAILED DESCRIPTION:
The limitations of the drugs used against HIV include their toxicity, their tolerability, their propensity to induce resistance when not taken with absolute regularity and their cost. Treatment interruption in patients receiving antiretroviral treatment in the setting of chronic infection is associated with viral rebound and rapid CD4 T cell decrease conducting to antiretroviral therapy restart. In patients with high CD4+ cell counts (patients receiving treatment of chronic infection with controlled viremia and patients who are receiving highly active antiretroviral therapy (HAART) now in whom treatment would not have been started based on current guidelines), the investigators evaluated whether the adjunctional of interferon alfa 2b to 3 structured treatment interruptions correlated with a long time off treatment. HAART was interrupted for 4 weeks, restarted and continued for 12 weeks. After 3 such cycles treatment was indefinitely suspended 48 weeks after study entry. Another aim of this study was to assess the immunological and virological factors associated with the duration of treatment interruption (proviral HIV DNA at baseline and during follow-up, plasma HIV RNA at baseline and during follow-up, CD4 T cell and CD8 T cell HIV specific responses at baseline and after 6 months of interruption).

ELIGIBILITY:
Inclusion Criteria:

* Males and non pregnant females
* Confirmed laboratory diagnosis of HIV infection
* Have been on the same continuous HAART regimen for at least 6 months prior to inclusion
* Viral load below 50 cp/ml for at least 6 months
* CD4 over 350 cells/mm3
* Previous viral load over 10000 cp/ml in their history
* No CD4 cell count under 100/mm3 in their history
* For women of reproductive ages: negative serum pregnancy test
* Signed written consent to participate.

Exclusion Criteria:

* Already had interferon or interleukin-2 (IL-2)
* Positive hepatitis C virus (HCV) PCR
* Under treatment with abacavir during screening
* Serious psychiatric history, suicide attempt, or severe depression
* History of thyroid abnormality
* Opportunistic infection ongoing
* Lymphoma or Kaposi's sarcoma (KS) under chemotherapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-12; Study Completion 2005-01

PRIMARY OUTCOMES:
Proportion of patients who did not reach the criteria to resume antiretroviral treatment at week 72 [W 72] (viral load over 30000 cp/ml at two consecutive monthly samples and/or CD4 count below 350/mm3 at two consecutive monthly samples)

SECONDARY OUTCOMES:
Viral rebound one and 3 months after stopping all antiviral treatments
Specific anti-HIV CD4 and CD8 response
Proviral HIV DNA at baseline and during follow-up
Description of genetic HIV viral mutations during procedure
Safety

CONTACTS AND LOCATIONS:
Overall Officials: François Boue, MD, Principal Investigator — Hopital Antoine Beclere service de Medecine Interne Clamart France; Dominique Costagliola, Study Chair — INSERM U 720
Locations (1):
- Service de Medecine Interne, Clamart, France